CLINICAL TRIAL: NCT00618943
Title: Treating Tobacco Dependence in Adolescents With Co-occurring Psychiatric Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jodi Prochaska, Associate Professor in Residence, University of California, San Francisco
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-09253; P50DA009253 (NIH)
Record Dates: First submitted 2008-02-15; First posted 2008-02-20 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Tobacco Use Cessation; Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

INTERVENTIONS:
Behavioral: Tobacco Use Cessation — The proposed intervention will proceed in three steps. Step 1, provided to all intervention participants, includes multimedia, stage-based, expert-system contacts at intake, 3- and 6-months follow-up supported with brief (15-min) motivational counseling sessions. Step 2, reserved for intervention participants interested in quitting, consists of 12-weeks of individual CBT sessions for smoking cessation. Step 3, a 12-week course of nicotine patch, will be offered to adolescents who enter the CBT Cessation Treatment, who do not have any medical contraindications, and who smoke an average of 5 cigarettes or more per day in the past month.

SUMMARY:
This research aims to identify efficacious strategies for treating tobacco dependence among adolescent smokers with co-occurring psychiatric disorders. Adolescent smoking remains a significant public health issue with 23% of high school students reporting smoking a cigarette in the past month1. Smoking rates are two to four times higher among adolescents with psychiatric disorders such as attention deficit disorders, conduct disorder, depression, anxiety disorders, and alcohol and illicit drug dependencies2-4.

Empirical investigations of adolescent tobacco treatment interventions number less than 50 with many of the studies criticized for methodological problems (i.e., follow up < 6 months, poor retention, lack of control or comparison groups)2,5, 6. There have been no unequivocal successes; however, promising interventions include stage-based, cognitive behavioral (CBT), and multicomponent treatments2, 7. Additionally, the nicotine patch is well tolerated and safe among adolescents8 and rarely abused9. Less than a third of adolescent tobacco users report intention to quit in the near future2, 10, 11; thus, it seems critical that cessation interventions for this complex group be designed to assist smokers at all stages of readiness through the quitting process. A stepped care approach has the potential of matching more intensive services to those ready for and in need of greater treatment. Interventions delivered in health care settings have the appeal of broad reach.

The primary specific aims of this research are to evaluate, in a randomized clinical trial (N=160), the efficacy of a stepped care intervention for treating smoking among adolescents recruited from outpatient psychiatry settings. To our knowledge, this would be the first study to examine outpatient psychiatry settings for treating tobacco dependence in adolescents. The stepped care intervention combines expert-system contacts, individual CBT sessions, and 12-weeks of nicotine replacement therapy (NRT).

ELIGIBILITY:
Inclusion Criteria:

* receiving active outpatient psychiatric care
* report smoking at least 1 cigarette in the previous 30 days and at least 100 cigarettes in their lifetime
* Other inclusion criteria are: no plan to relocate outside of the greater San Francisco Bay Area in the next 12 months and telephone access for scheduling follow up assessments.

Exclusion Criteria:

* cognitive impairment precluding ability to participate
* non-English speaking
* currently engaged in tobacco treatment
* Recruitment of acutely psychotic, manic, or hostile patients will be delayed until there is significant reduction of these symptoms and patients are able to assent to study participation

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
7 day point prevalence of cigarette abstinence | 3, 6, 12 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Judith J Prochaska, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Edgewood Center for Children and Families, San Bruno, California
  - UCSF Langley Porter Psychiatric Institute, San Francisco, California
  - San Mateo County Mental Health, San Mateo, California